CLINICAL TRIAL: NCT00004001
Title: Docetaxel and Estramustine Versus Mitoxantrone and Prednisone for Advanced, Hormone Refractory Prostate Cancer
Brief Title: S9916, Combination Therapy in Treating Patients With Advanced Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067211; S9916 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Mitoxantrone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel and Estramustine (Experimental): Estramustine, 280 mg, PO, TID, Days 1-5; q 21 days Docetaxel, 60mg/m2, IV, Day 2; q 21 days
  Interventions: Drug: docetaxel; Drug: estramustine
- Mitoxantrone and Prednisone (Active Comparator): Mitoxantrone, 12 mg/m2, IV, Day 1; q 21 days Prednisone, 5 mg, PO, BID, Days 1-21; q 21 days
  Interventions: Drug: mitoxantrone; Drug: prednisone

INTERVENTIONS:
Drug: docetaxel
  Arms: Docetaxel and Estramustine
Drug: estramustine
  Arms: Docetaxel and Estramustine
Drug: mitoxantrone
  Arms: Mitoxantrone and Prednisone
Drug: prednisone
  Arms: Mitoxantrone and Prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy and hormone therapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells. It is not yet known whether estramustine plus docetaxel is more effective than mitoxantrone plus prednisone for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of estramustine plus docetaxel with that of mitoxantrone plus prednisone in treating patients who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and progression-free survival in patients with hormone-refractory, metastatic adenocarcinoma of the prostate treated with docetaxel and estramustine vs mitoxantrone and prednisone.
* Compare the qualitative and quantitative toxic effects of these regimens in this patient population.
* Compare the quality of life, including palliation of metastatic bone pain and global quality of life, of patients treated with these regimens.
* Record prostate-specific antigen values for future correlations with response and survival in patients treated with these regimens.
* Compare the responses in patients with bidimensionally measurable disease treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease status (measurable or evaluable disease progression vs rising PSA only), NCI Common Toxicity Criteria version 2.X pain scale (grade 2 or greater vs less than 2), and SWOG performance status (0-1 vs 2-3). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV over 1 hour on day 2.
* Arm II: Patients receive mitoxantrone IV over 30 minutes on day 1 and oral prednisone twice daily on days 1-21.

Treatment in both arms repeats every 3 weeks for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.

Quality of life is assessed at baseline, after courses 4 and 8, and then at 1 year after randomization.

Patients are followed every 6 months for 2 years and then annually for 1 year.

PROJECTED ACCRUAL: A total of 620 patients (310 per arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the prostate
* Unresponsive or refractory to hormonal therapy, as defined by at least 1 of the following criteria:

  * Progression of bidimensionally measurable disease
  * Progression of evaluable but not measurable disease (bone scan)
  * At least 2 consecutive rises in PSA and a PSA level of at least 5 ng/mL
* No minimum PSA required for measurable disease or non-PSA evaluable disease
* Soft tissue disease that has been irradiated within the past 2 months is not considered measurable disease
* Prior orchiectomy OR
* Medical castration using leuprolide or goserelin

  * Luteinizing hormone-releasing hormone (LHRH) agonist therapy must continue during study
* Prior nonsteroidal antiandrogens (flutamide, ketoconazole, bicalutamide, or nilutamide) allowed if disease progression occurred
* No third-space fluid accumulation such as ascites or symptomatic pleural effusion
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-3
* Performance status 3 must be due to pain secondary to bone metastases

Life expectancy:

* Not specified

Hematopoietic:

* No hypercoagulability

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No history of myocardial infarction
* No history of congestive heart failure unless well controlled
* No history of cerebrovascular accident or atrial fibrillation
* No active thrombophlebitis
* Left ventricular ejection fraction (LVEF) at least 50% by Multi Gated Acquisition Scan (MUGA) scan or 2-D echocardiogram

Pulmonary:

* No history of pulmonary embolus

Other:

* Recovered from major infections
* No other significant active medical illness
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No more than 1 prior biologic therapy regimen
* No concurrent biological response modifiers

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered
* No more than 1 prior chemotherapy regimen
* No prior estramustine, taxanes, anthracyclines, or mitoxantrone
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior flutamide or ketoconazole (6 weeks for bicalutamide or nilutamide)
* No concurrent corticosteroids or hormonal therapy (except megestrol for hot flashes or continuing LHRH treatment)

Radiotherapy:

* See Disease Characteristics
* Prior samarium Sm 153 lexidronam pentasodium allowed
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to 30% or more of bone marrow
* No prior strontium chloride Sr 89
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior surgery and recovered

Other:

* At least 4 weeks since prior bisphosphonates
* No prior anticoagulation therapy (i.e., warfarin), except aspirin
* No concurrent bisphosphonates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 1999-10; Primary Completion 2006-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Compare overall survival in the two study arms | up to 4 years
  Measured from date of registration to date of death due to any cause

SECONDARY OUTCOMES:
Compare progression-free survival between two study arms | up to 4 years
  Measured from date of registration to date of first observation of progression disease, or death due to any cause
Compare Prostate-Specific Antigen (PSA) response between two study arms | up to 4 years or time of disease progression
  A confirmed partial response of non-measurable disease was defined as a reduction by more than 50% over baseline in two or more Prostate-Specific Antigen (PSA) measurements obtained at least four weeks apart, with no evidence of disease progression on imaging. Progressive disease was defined as a 25% increase in the serum PSA level - to at least 5 ng per milliliter - over the last preregistration measurement, with confirmation of the increase at least four weeks later. For patients with a decrease in serum PSA levels during the trial, progressive disease was defined as a confirmed increase of 25%, to at least 5 ng per milliliter over the nadir.
Compare objective responses between two study arms | up to 12 cycles of treatment ( 1cycle = 21 days)
  Objective responses were defined on the basis of the sum of bi-dimensional measurements of metastatic lesions. Confirmed objective responses required a follow-up scan (a minimum of four weeks later) that demonstrated a continued response. Progression was defined by one of the following: a 50 percent increase or an increase of 10 cm^2, whichever was smaller, in the sum of measurements of metastatic lesions over the sum at baseline; a clear worsening of nonmeasurable disease; reappearance of any lesion that had disappeared; appearance of any new lesion; or death.
Compare toxicities between the two study arms | up to 12 cycles of treatment (1 cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P. Petrylak, MD, Study Chair — Herbert Irving Comprehensive Cancer Center; Eric J. Small, MD, Study Chair — University of California, San Francisco; Patrick A. Burch, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health System, Grand Forks, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] Hussain M, Goldman B, Tangen C, Higano CS, Petrylak DP, Wilding G, Akdas AM, Small EJ, Donnelly BJ, Sundram SK, Burch PA, Dipaola RS, Crawford ED. Prostate-specific antigen progression predicts overall survival in patients with metastatic prostate cancer: data from Southwest Oncology Group Trials 9346 (Intergroup Study 0162) and 9916. J Clin Oncol. 2009 May 20;27(15):2450-6. doi: 10.1200/JCO.2008.19.9810. Epub 2009 Apr 20. PMID 19380444
- [Background] de Wit R. Chemotherapy in hormone-refractory prostate cancer. BJU Int. 2008 Mar;101 Suppl 2:11-5. doi: 10.1111/j.1464-410X.2007.07485.x. PMID 18307687
- [Background] Goldman B, Hussain M, Tangen C, et al.: Prostate-specific antigen progression (PSA-P) as a predictor of overall survival (OS) in patients (pts) with metastatic prostate cancer (PC): data from S9346 and S9916. [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-165, 2008.
- [Background] Hussain MH, Goldman B, Tangen CM, et al.: Use of prostate-specific antigen progression (PSA-P) to predict overall survival (OS) in patients (pts) with metastatic prostate cancer (PC): data from S9346 and S9916. [Abstract] J Clin Oncol 26 (Suppl 15): A-5015, 2008.
- [Background] Calabro F, Sternberg CN. Current indications for chemotherapy in prostate cancer patients. Eur Urol. 2007 Jan;51(1):17-26. doi: 10.1016/j.eururo.2006.08.013. Epub 2006 Aug 22. PMID 17007996
- [Background] Chowdhury S, Burbridge S, Harper PG. Chemotherapy for the treatment of hormone-refractory prostate cancer. Int J Clin Pract. 2007 Dec;61(12):2064-70. doi: 10.1111/j.1742-1241.2007.01551.x. Epub 2007 Oct 23. PMID 17956560
- [Background] Mendiratta P, Armstrong AJ, George DJ. Current standard and investigational approaches to the management of hormone-refractory prostate cancer. Rev Urol. 2007;9 Suppl 1(Suppl 1):S9-S19. PMID 17387372
- [Background] Montgomery RB, Goldman B, Tangen CM, Hussain M, Petrylak DP, Page S, Klein EA, Crawford ED; Southwest Oncology Group. Association of body mass index with response and survival in men with metastatic prostate cancer: Southwest Oncology Group trials 8894 and 9916. J Urol. 2007 Nov;178(5):1946-51; discussion 1951. doi: 10.1016/j.juro.2007.07.026. Epub 2007 Sep 17. PMID 17868721
- [Background] Burgess EF, Roth BJ. Changing perspectives of the role of chemotherapy in advanced prostate cancer. Urol Clin North Am. 2006 May;33(2):227-36, vii. doi: 10.1016/j.ucl.2005.12.006. PMID 16631461
- [Background] Lucas A, Petrylak DP. The case for early chemotherapy for the treatment of metastatic disease. J Urol. 2006 Dec;176(6 Pt 2):S72-5. doi: 10.1016/j.juro.2006.06.077. PMID 17084173
- [Background] Moss RA, Petrylak DP. Cytotoxic chemotherapy for prostate cancer: Who and when? Curr Treat Options Oncol. 2006 Sep;7(5):370-7. doi: 10.1007/s11864-006-0005-x. PMID 16904054
- [Background] McKeage K, Keam SJ. Docetaxel in hormone-refractory metastatic prostate cancer. Drugs. 2005;65(16):2287-94; discussion 2295-7. doi: 10.2165/00003495-200565160-00003. PMID 16266195
- [Result] Moinpour CM, Donaldson GW, Nakamura Y. Chemotherapeutic impact on pain and global health-related quality of life in hormone-refractory prostate cancer: Dynamically Modified Outcomes (DYNAMO) analysis of a randomized controlled trial. Qual Life Res. 2009 Mar;18(2):147-55. doi: 10.1007/s11136-008-9433-3. Epub 2009 Jan 9. PMID 19130298
- [Result] Petrylak DP, Ankerst DP, Jiang CS, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Evaluation of prostate-specific antigen declines for surrogacy in patients treated on SWOG 99-16. J Natl Cancer Inst. 2006 Apr 19;98(8):516-21. doi: 10.1093/jnci/djj129. PMID 16622120
- [Result] Southwest Oncology Group; Berry DL, Moinpour CM, Jiang CS, Ankerst DP, Petrylak DP, Vinson LV, Lara PN, Jones S, Taplin ME, Burch PA, Hussain MH, Crawford ED. Quality of life and pain in advanced stage prostate cancer: results of a Southwest Oncology Group randomized trial comparing docetaxel and estramustine to mitoxantrone and prednisone. J Clin Oncol. 2006 Jun 20;24(18):2828-35. doi: 10.1200/JCO.2005.04.8207. PMID 16782921
- [Result] Berry DL, Moinpour CM, Jiang C, et al.: Quality of life (QOL) and pain in advanced stage prostate cancer: impact of missing data on evaluating palliation in SWOG 9916. [Abstract] J Clin Oncol 22 (Suppl 14): A-4579, 401s, 2004.
- [Result] Crawford ED, Pauler DK, Tangen CM, et al.: Three-month change in PSA as a surrogate endpoint for mortality in advanced hormone-refractory prostate cancer (HRPC): data from Southwest Oncology Group study S9916. [Abstract] J Clin Oncol 22 (Suppl 14): A-4505, 383s, 2004.
- [Result] Petrylak DP, Tangen C, Hussain M, et al.: SWOG 99-16: randomized phase III trial of docetaxel (D)/estramustine (E) versus mitoxantrone(M)/prednisone(p) in men with androgen-independent prostate cancer (AIPCA). [Abstract] J Clin Oncol 22 (Suppl 14): A-3, 2s, 2004.
- [Result] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Result] Hussain M, Petrylak D, Fisher E, Tangen C, Crawford D. Docetaxel (Taxotere) and estramustine versus mitoxantrone and prednisone for hormone-refractory prostate cancer: scientific basis and design of Southwest Oncology Group Study 9916. Semin Oncol. 1999 Oct;26(5 Suppl 17):55-60. PMID 10604271
- [Derived] Unger JM, LeBlanc M, Blanke CD. The Effect of Positive SWOG Treatment Trials on Survival of Patients With Cancer in the US Population. JAMA Oncol. 2017 Oct 1;3(10):1345-1351. doi: 10.1001/jamaoncol.2017.0762. PMID 28586789